CLINICAL TRIAL: NCT04928664
Title: Continuous Standard Bupivacaine Versus Single Liposomal Bupivacaine Injection for Interscalene Brachial Plexus Block for Pain Management After Proximal Humerus Fracture Fixation
Brief Title: Continuous vs Liposomal Bupivacaine Interscalene Block for Proximal Humeral Fracture (CLIP)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chan Chi-Wing, Honorary Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 20-247
Record Dates: First submitted 2021-06-01; First posted 2021-06-16 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Shoulder Fractures
Keywords: liposomal bupivacaine; interscalene block
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Intervention Model Description: A separate anaesthetist will then prepare 10 ml of LB or SB, and a covered elastomeric pump that is either filled with 300ml NS or with 300ml 0.2% SB according to the group assigned for the attending anaesthetist.
Who Masked: Participant, Investigator
Masking Description: The subjects, the investigators, and all the parties involved in patient management or data collection will be blinded throughout the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liposoaml Bupivacaine (LB) Group (Active Comparator): Intervention group
  Interventions: Drug: Liposomal bupivacaine
- Standard Bupivacaine (SB) Group (Experimental): Control group
  Interventions: Drug: Standard bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — Single shot injection of 10ml 1.33% LB; Due to the milky colour of LB, syringe containing the LB will be covered; Followed by placement of indwelling catheter in ISB; Catheter will be connected to a fixed-rate portable elastometric pump ( Easy pump, ®) upon arrival in the recovery room by the nurse; The pump will be filled with 300ml NS; The default fixed rate of infusion will be 5ml/hr; Both the pump and the clamp will be covered by an aluminium foil; Catheter and pump will be removed on post-operative day 2
  Arms: Liposoaml Bupivacaine (LB) Group
Drug: Standard bupivacaine — Single shot injection of 10 ml 0.25% SB in ISB; In order to have blinding to the drug injected, syringe containing SB will be covered; followed by placement of indwelling catheter in ISB; Catheter will be connected to a fixed-rate portable elastometric pump ( Easy pump, ®) upon arrival in the recovery room by the nurse; The pump will be filled with 300ml 0.2% SB; The default fixed-rate of infusion will be 5ml/hr; Both the pump and the clamp will be covered by an aluminium foil; Catheter and pump will be removed on post-operative day 2
  Arms: Standard Bupivacaine (SB) Group

SUMMARY:
Restricted range of shoulder motion following ORIF is a potential complication that severely affects the patients' functional outcome and should be actively avoided by means of adequate pain control in addition to early mobilization and physiotherapy.

Peripheral nerve blocks, which can be given as a single injection or continuous infusion via an indwelling catheter, are analgesic options to be considered. Interscalene Block (ISB) is the regional analgesia of choice for the shoulder and proximal humerus region. While continuous infusion (aka continuous nerve block) offers the advantage of a longer duration of analgesia compared to a single injection of standard local anaesthetic, it is associated with an inherent risk of catheter displacement, dislodgement, obstruction, and infection.

Compared to Standard Bupivacaine (SB), Liposomal Bupivacaine (LB) is a formulation designed to prolong the duration of action to up to 72 hours by slow release of bupivacaine from the multi-vesicular liposomes. Several studies have demonstrated satisfactory analgesic effects of liposomal bupivacaine given as local surgical site infiltration over placebo. However, the effects of single injection of liposomal bupivacaine given via local surgical site infiltration compared to continuous nerve block have been inconsistent. Administrating liposomal bupivacaine directly to peripheral nerve blocks is a potentially effective approach that has not been extensively studied. ISB with single shot liposomal bupivacaine has been shown to provide superior postoperative analgesia compared to ISB with injection of standard bupivacaine or placebo. ISB with liposomal bupivacaine could perhaps prolong and improve postoperative analgesia without the potential problems with continuous nerve blocks. The analgesic effect of ISB with single shot liposomal bupivacaine versus continuous ISB with standard bupivacaine has not been previously investigated. The aim of this study is to compare the analgesic effect of these two analgesic modalities for plate fixation of proximal humerus fractures.

DETAILED DESCRIPTION:
CONDUCT OF ISB:

Side effects and potential complications will be explained and informed consent will be obtained from all subjects.

Time-out will be performed before the start of ISB in accordance with the WHO checklist, confirming the side of surgery with the subject.

Standard monitoring will be placed and an intravenous catheter will be established.

All ISB will be performed by anaesthetists experienced in ultrasound-guided ISB.

An aseptic technique will be applied. ISB will be performed under ultrasound guidance in an in-plane manner. Catheter-over-needle set with a 50mm short-bevel insulated needle will be used.

Placement of needle will be confirmed with sonoanatomy, absence of persistent paraesthesia, negative aspiration of air and blood, real-time visualisation of the spread of drug and low resistance upon injection. The catheter will be left in-situ and sutured to the skin after injection of the drug and withdrawal of the needle.

Neither the supraclavicular nerve nor the suprascapular nerve will be blocked.

The use of a peripheral nerve stimulator and administration of sedation will be at the discretion of the attending anaesthetist.

A successful ISB is defined as loss of cold sensation to ice in the C5 dermatome, which will be tested by the attending anaesthetist in addition to assessing the presence of aforementioned complications before induction of general anaesthesia.

ANAESTHESIA & ANALGESIA:

(I) PRE-OPERATIVE:

Routine preoperative assessment will be taken at the pre-admission clinic or at the general ward, followed by these orders:

ECG and chest x-ray Standard fasting times (6 hours for solid food and 2 hours for clear liquid) No analgesics or sedatives as premeditation

(II) INTRA-OPERATIVE: ISB will be performed as described above before induction of General Anaesthesia (GA).

For Induction of GA:

IV Fentanyl 1-2mcg/kg IV Propofol 2-4 mg/kg IV Rocuronium 0.6-1mg/kg

For Maintenance of GA:

Target controlled infusion of propofol at an effect site concentration of 0-1.5 mcg/ml Air/O2/desflurane, target MAC: 0.6 -1.0 IV Morphine 3mg before skin incision IV Remifentanil 0.1-0.2 mcg/kg/min, target SBP not more than 20% increase from baseline Choice of muscle relaxant and IV fluid at the discretion of the attending anaesthetist Vasopressors, anti-hypertensive medications, anti-arrhythmia medications may be given as necessary No Paracetamol / NSAID / Ketamine / Dexmedetomidine / IV Lidocaine infusion / Magnesium No LA infiltration

For Emergence from GA:

IV Ondansetron 4mg 30 minutes before the end of surgery Reversal will be achieved with 2.5 mg of neostigmine and 1.2 mg of atropine and patients will be extubated when ventilation and consciousness is adequate

(III) POST-OPERATIVE (RECOVERY IN PACU): All subjects will be transferred to PACU for further monitoring for at least 30 minutes.

The indwelling catheter will be connected to a fixed-rate portable elastometric pump ( Easy pump, ®) upon arrival in the recovery room by the nurse.

Pain at rest will be evaluated every 5 mins using NRS. If the score is greater than 4/10, 2mg morphine will be given intravenously every 5 mins provided the subject has a respiratory rate of > 12/min and a sedation score of <1 until a NRS of < 4/10 is achieved.

The presence of complications will be assessed by the attending anaesthetist before discharge from PACU.

(IV) POST-OPERATIVE (IN WARD): BP, heart rate, SpO2, and sedation score will be monitored at 1-hour intervals while on PCA morphine; BP and heart rate will be monitored at 4-hour intervals once PCA morphine is terminated.

Diet will be resumed on Post-Operative Day 0. All subjects will undergo standard institutional rehabilitation program, which consists of supervised passive forward flexion and external rotation exercise for 3 weeks, followed by assisted active movements till 6 weeks.

Standardized analgesic regime will be prescribed:

IV PCA morphine for 2 days PO paracetamol 500mg QID for 2 weeks PO celecoxib 200mg daily for 3 days IMI morphine 0.1mg/kg Q4H prn as rescue analgesic for 3 days IV ondansetron 0.1mg/kg Q8H prn for 3 days PO Dihydrocodeine 30mg TDS prn from POD3 to PO7

Signs and symptoms of complications will be assessed by the pain team daily until postoperative day 2 when the pump and catheter will be removed. Pain assessment and side effects related to analgesic will be assessed by the pain team daily until postoperative day 2, followed by phone follow-up until postoperative day 7

For phone follow-up, patients will be received a phone call in the afternoon at around 3 pm for both pain score and Overall Benefit of Analgesic Scale (OBAS)

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Age between 18 and 80
* Proximal humeral fracture

Exclusion Criteria:

* Surgical exclusion criteria:
* Revision surgery
* Pathological fracture
* 4-part or shaft fracture
* Multiple fractures
* Unable to attend rehabilitation
* Preexisting shoulder problems
* Abbreviated Mental Test Score (AMT score) < 8
* Allergy to amide local anaesthetics, paracetamol, non-steroidal anti-inflammatory drugs (NSAIDS), opioids
* Respiratory Disease with limited respiratory reserve
* Cardiac Disease: Any degree of Heart Block, Heart Failure
* Neurological: Any Seizure Disorder
* Psychiatric illnesses affecting pain perception e.g. severe depression and anxiety disorder
* Alcohol or substance abuse
* Chronic Pain, other than chronic knee pain
* Daily use of strong opioids (morphine, fentanyl, hydromorphone, ketobemidone, methadone, diamorphine, oxycodone, or meperidine) before operation
* Impaired Renal Function (defined as preoperative eGFR < 30ml /min /1.73 m2)
* Impaired Hepatic Function
* Pregnancy
* Inability to use PCA
* Patient refusal to ISB
* Patient refusal to study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2019-06-04 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Numerical Rating Score (NRS) | Changes from baseline NRS at day 7
  NRS (movement) = NRS during attempted passive forward flexion to 90 degrees NRS (rest) = NRS at rest
  Pain at rest will be evaluated every 5 mins using NRS during recovery in PACU. NRS ranges from 0 to 10, where 0= no pain and 10= the worst imageable pain

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - The University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No